CLINICAL TRIAL: NCT01228058
Title: A Prospective Evaluation of Thromboelastography for Identifying Coagulopathy in Severely Injured Patients
Acronym: RapidTEG
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Haemonetics Corporation (Industry)
Responsible Party: Principal Investigator, Bryan Cotton, Visiting Associate Professor - Surgery, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-10-0160
Record Dates: First submitted 2010-10-20; First posted 2010-10-25 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Coagulopathy
Keywords: Trauma; Coagulopathy; Coagulopathy in adult trauma patients
MeSH Terms: conditions — Hemostatic Disorders; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult trauma patients: Patients admitted to the emergency department (ED) as the highest level of acuity following a traumatic injury at three Level 1 trauma centers in the United States (UT Houston, UC San Francisco, Oregon Health Center).
  Interventions: Procedure: RapidTEG test

INTERVENTIONS:
Procedure: RapidTEG test — The RapidTEG test will be done at the study time points (3, 6, 12, 24 hours and 4 addiitonal days).

SUMMARY:
The purpose of this study is to evaluate the clinical utility of thrombelastography (TEG) to predict and identify trauma patients at increased risk of receiving blood transfusion, develop multiple organ failure and mortality.

TEG has been proposed as a superior tool to rapidly diagnose and help guide resuscitation with blood products and preclinical data suggest that TEG is both more sensitive and specific than PT or PTT for coagulation abnormalities. Based on the preclinical work led by Dr. Holcomb, our hypothesis is that the Rapid TEG will help to identify these coagulopathic patients earlier, allow for rapid MT protocol activation, and assist in developing data driven blood product transfusion guidelines.

DETAILED DESCRIPTION:
This protocol is based on the fact that approximately 30% of severely injured military and civilian patients have disturbances of coagulation immediately upon arrival to the trauma center by traditional coagulation testing. It is hypothesized that:

1. the coagulopathy of these patients may be detected more rapidly with RapidTEG than with traditional coagulation testing (prothrombin time, PT; international normalized ratio, INR; activated partial thromboplastin time, aPTT).
2. the disturbances in the different RapidTEG parameters will correlate with early blood product utilization.
3. the RapidTEG parameters will correlate closely with patient outcomes.
4. the Rapid TEG will be able to describe the changes that occur with coagulation over time and do so for patients with different injury mechanisms and severities

This group has recently completed enrollment on the PRospective, Observational, Multi-center Massive Transfusion sTudy (PROMMTT) to evaluate the process, the decision-making, and outcomes associated with MT. This trial is supported by a ten million dollar grant from the U.S. Department of Defense for the Center for Translational Injury Research (CeTIR) and it investigators to conduct a multi-site observational study of severely injured trauma patients who require blood transfusions. Through our efforts, we hope to determine the best method of identifying patients who will benefit from receiving different ratios of red blood cells to plasma to platelets. This study was also designed to evaluate existing MT protocols at ten leading trauma centers and to identify which protocols are associated with better survival. Results of this study will be used to develop a future randomized clinical trial that will test these protocols.

Building on the authors proven experience with (1) predictive scoring methods to predict massive transfusion, (2) creation and maturation of a massive transfusion protocol, and (3) design of large, multi-institutional studies, the PROMMTT investigators will conduct a prospective cohort study of severely injured patients (major trauma activations) arriving to three ACS-verified academic Level 1 Trauma Centers, in which the following 3 aims will be addressed:

1. To determine the prevalence and severity of immediate disturbances in coagulation by both RapidTEG and conventional coagulation parameters among major trauma activations.
2. To determine if there are specific abnormalities of RapidTEG that correlate with specific early blood product utilization.
3. To determine if RapidTEG abnormalities, when compared to kaolin-activated TEG, PT, INR and aPTT, correlate with patient outcomes in severely injured patients.
4. To determine the temporal relationship between RapidTEG parameters and anatomic injury, mechanism of injury, and severity of injury.

TEG has been proposed as a superior tool to rapidly diagnose and help guide resuscitation with blood products and preclinical data suggest that TEG is both more sensitive and specific than PT or PTT for coagulation abnormalities. Based on the preclinical work led by Dr Holcomb, we feel that the Rapid TEG will help to identify these coagulopathic patients earlier, allow for rapid MT protocol activation, and assist in developing data driven blood product transfusion guidelines. While the TEG machine is not new, widespread and thoughtful implementation in the trauma arena has not occurred. There are no transfusion algorithms constructed on large numbers of patients, admission TEG and PT/PTT values, transfusion amounts and patient outcomes. We feel that a logical step-by-step program that first constructs a data driven algorithm, and then validates the algorithm is the safest pathway to follow.

We plan to perform RapidTEG upon admission, at 3-hours post-admission, 6-hours post-admission, 12-hours post-admission, 24-hours post-admission, and then daily for 4 additional days. Blood samples (2 mL non-citrated fresh whole blood) will be obtained in addition to standard blood samples for major trauma patients. RapidTEG will be performed using the Thrombelastograph 5000 (Hemoscope Corporation, Niles, IL). Coagulation will be activated by tissue factor. Standard parameters will be obtained using Hemoscope software: TEG-ACT, r-time, K-time, alpha angle, maximum amplitude (mA), and LY30. In addition to RapidTEG, we plan to perform conventional kaolin-activated TEG, prothrombin time (PT), international normalized ratio (INR), activated thromboplastin time (aPTT), and platelet count using standard methods. The time from obtaining the blood sample until the time that the results are made available will also be recorded for all parameters tested. For the RapidTEG, this will include the final results for the test as well as the times that the TEG-ACT, alpha angle, and MA become available by graphical display.

ELIGIBILITY:
Inclusion Criteria:

* Major trauma patients who require the highest level of trauma team activation at each site.
* Estimated age of 18 or higher
* Transfers less than 6 hours post-injury Exclusion Criteria: -Children less than 18 years of age.
* Burns > 20% of body surface area
* CPR pre-hospital
* Prisoners - defined as anyone directly admitted from a correctional facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is all major-trauma patients admitted to one of the three participating ACS-verified academic Level 1 trauma centers.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and severity of immediate disturbances in coagulation by both RapidTEG and conventional coagulation parameters among major trauma activations. | First 5 days of hospitalization

SECONDARY OUTCOMES:
To determine if there are specific abnormalities of RapidTEG that correlate with specific early blood product utilization. | First 5 days of hospitalization
To determine if RapidTEG abnormalities, when compared to kaolin-activated TEG, PT, INR and aPTT, correlate with patient outcomes in severely injured patients. | First 5 days of hospitalization
To determine the temporal relationship between rapid TEG parameters and anatomic injury, mechanism of injury, and severity of injury. | First 5 days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Cotton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - University of California - San Francisco, San Francisco, California
  - Oregon Health and Science University, Portland, Oregon
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas

REFERENCES:
- [Background] Acosta JA, Yang JC, Winchell RJ, Simons RK, Fortlage DA, Hollingsworth-Fridlund P, Hoyt DB. Lethal injuries and time to death in a level I trauma center. J Am Coll Surg. 1998 May;186(5):528-33. doi: 10.1016/s1072-7515(98)00082-9. PMID 9583692
- [Background] Brohi K, Singh J, Heron M, Coats T. Acute traumatic coagulopathy. J Trauma. 2003 Jun;54(6):1127-30. doi: 10.1097/01.TA.0000069184.82147.06. PMID 12813333
- [Background] Cotton BA, Gunter OL, Isbell J, Au BK, Robertson AM, Morris JA Jr, St Jacques P, Young PP. Damage control hematology: the impact of a trauma exsanguination protocol on survival and blood product utilization. J Trauma. 2008 May;64(5):1177-82; discussion 1182-3. doi: 10.1097/TA.0b013e31816c5c80. PMID 18469638
- [Background] Niles SE, McLaughlin DF, Perkins JG, Wade CE, Li Y, Spinella PC, Holcomb JB. Increased mortality associated with the early coagulopathy of trauma in combat casualties. J Trauma. 2008 Jun;64(6):1459-63; discussion 1463-5. doi: 10.1097/TA.0b013e318174e8bc. PMID 18545109
- [Background] MacLeod JB, Lynn M, McKenney MG, Cohn SM, Murtha M. Early coagulopathy predicts mortality in trauma. J Trauma. 2003 Jul;55(1):39-44. doi: 10.1097/01.TA.0000075338.21177.EF. PMID 12855879
- [Background] Cotton BA, Au BK, Nunez TC, Gunter OL, Robertson AM, Young PP. Predefined massive transfusion protocols are associated with a reduction in organ failure and postinjury complications. J Trauma. 2009 Jan;66(1):41-8; discussion 48-9. doi: 10.1097/TA.0b013e31819313bb. PMID 19131804